CLINICAL TRIAL: NCT03016741
Title: Cognitive Effects of Androgen Receptor (AR) Directed Therapies for Advanced Prostate Cancer
Brief Title: Cognitive Effects of Androgen Receptor Directed Therapies for Advanced Prostate Cancer
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 17U19; STU00206082 (Registry Identifier: Northwestern University); NCI-2016-01795 (Other: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2016-12-01; First posted 2017-01-11 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Castration-Resistant Prostatic Cancer; Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer; Hormone-Refractory Prostate Cancer
Keywords: cognitive function; hormonal therapy; cancer survivorship; dementia; cognitive dysfunction; mild cognitive impairment
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms; Dementia; Cognitive Dysfunction | interventions — Gonadotropin-Releasing Hormone; Prednisone; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (abiraterone acetate, prednisone) (Other): Patients receive standard of care treatment with GnRH agonist/antagonist therapy. Patients also receive abiraterone acetate PO and prednisone PO BID in the absence of disease progression or unacceptable toxicity. Patients then undergo cognitive assessment comprising of neuro-cognitive tests and assessments of overall quality of life, fatigue, pain, and symptoms at baseline, 3, 6, and 12 months. Patients also undergo MRI program for 40 minutes comprising of DTI, fMRI, ASL MRI, MPRAGE MRI, FLAIR MRI, and BOLD MRI at baseline and 3 months.
  Interventions: Biological: GnRH agonist/antagonist; Drug: Prednisone; Drug: Abiraterone Acetate
- Arm II (enzalutamide) (Other): Patients receive standard of care treatment with GnRH agonist/antagonist therapy. Patients also receive enzalutamide PO QD in the absence of disease progression or unacceptable toxicity. Patients undergo cognitive assessment and MRI program as in Arm I.
  Interventions: Biological: GnRH agonist/antagonist; Drug: Enzalutamide

INTERVENTIONS:
Biological: GnRH agonist/antagonist — Given GnRH agonist/antagonist therapy
Drug: Prednisone — Given by mouth
  Arms: Arm I (abiraterone acetate, prednisone)
Drug: Abiraterone Acetate — Given by mouth
  Other Names: Zytiga
  Arms: Arm I (abiraterone acetate, prednisone)
Drug: Enzalutamide — Given by mouth
  Other Names: Xtandi
  Arms: Arm II (enzalutamide)

SUMMARY:
This clinical trial studies cognitive function in men with prostate cancer treated with androgen receptor directed therapies such as abiraterone acetate and enzalutamide. The investigators use MRI imaging (non-invasive, non-contrast) to see whether there are changes in brain structure or activity related to treatment that may be related to changes in cognitive function. The investigators are also looking for genetic variations that might make patients more or less sensitive to cognitive changes during treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare cognitive function and associated mediators of cognitive function (quality of life, depression, pain, and fatigue) of men with metastatic castration-resistant prostate cancer (mCRPC) or metastatic hormone sensitive prostate cancer during treatment with enzalutamide (mCRPC only) and abiraterone acetate (mHSPC or mCRPC).

SECONDARY OBJECTIVES:

I. To identify characteristics of men with mCRPC associated with change in cognitive function during treatment with androgen receptor (AR) directed therapy.

II. To compare quality of life and associated factors, including fatigue, pain, and depression, of men with mCRPC during treatment with enzalutamide and abiraterone acetate.

TERTIARY OBJECTIVES:

I. To analyze whether single nucleotide polymorphisms (SNPs) may be associated with change in cognitive function during treatment with AR directed therapy.

II. To compare the functional and structural components of the brain over time and between the brains of men with mCRPC treated with enzalutamide or abiraterone acetate using diffusion tensor imaging (DTI), functional MRI (fMRI), arterial spin labeling (ASL), and other advanced neuroimaging techniques.

OUTLINE: Treatment patients with metastatic castration-resistant prostate cancer are randomized to 1 of 2 arms. Control patients receiving long term androgen deprivation therapy will be assessed with the same measures as a control arm.

ARM I: Patients receive standard of care treatment with gonadotrophin releasing hormone (GnRH) agonist/antagonist therapy. Patients also receive abiraterone acetate orally (PO) and prednisone PO twice daily (BID) in the absence of disease progression or unacceptable toxicity. Patients then undergo cognitive assessment comprising of neuro-cognitive tests and assessments of overall quality of life, fatigue, pain, and symptoms at baseline, 3, 6, and 12 months. Patients also undergo MRI program for 40 minutes comprising of DTI, fMRI, ASL MRI, Magnetization Prepared Rapid Gradient Echo (MPRAGE) MRI, Fluid attenuated Inversion Recovery (FLAIR) MRI, and blood oxygenation level-dependent (BOLD) MRI at baseline and 3 months.

ARM II: Patients receive standard of care treatment with GnRH agonist/antagonist therapy. Patients also receive enzalutamide PO QD in the absence of disease progression or unacceptable toxicity. Patients undergo cognitive assessment and MRI program as in Arm I.

ARM III: Patients receive standard of care treatment with GnRH agonist/antagonist therapy and undergo cognitive assessment and MRI program as in Arm I.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of prostate cancer and have received treatment with GnRH agonist or antagonist therapy for at least 1 month prior to enrollment.
* Willing and able to complete survey questionnaires in English without assistance through the duration of the study. This stipulation is in place because not all of the proposed quality of life or cognitive tests are available or validated in other languages.
* Age ≥ 18 years.
* Ability to understand and the willingness to sign a written informed consent document written in English that is approved by an institutional review board.
* Have either newly diagnosed metastatic hormone sensitive prostate cancer (mHSPC) or castration-resistant metastatic prostate cancer (mCRPC) and eligible to undergo treatment with abiraterone acetate (mHSPC or mCRPC) or enzalutamide (mCRPC)
* Patients may have received the following prior AR directed therapy prior to enrollment: bicalutamide, ketoconazole. Prior to enrollment, patients may have received treatment with abiraterone acetate or enzalutamide for no more than 14 days before completing baseline studies.
* Patients may have received chemotherapy for hormone-sensitive metastatic prostate cancer only, but it must not have lasted for more than 6 months. At least 12 months must have elapsed since completion of chemotherapy.
* Patients may have received prior definitive radiation therapy or surgery. At least 60 days must have elapsed since completion of definitive radiation therapy or surgery and patient must have only grade 2 or less adverse effects at the time of registration. Enrollment during palliative radiation of ≤ 10 days, or radiation of ≤ 10 days during the duration of the study is allowed.
* Patients must be able to take oral medication.

Exclusion Criteria:

* Prior treatment with enzalutamide or abiraterone acetate for > 14 days prior to enrollment and completion of baseline tests.
* Receipt of chemotherapy for prostate or other cancer within the past 12 months with residual cognitive deficits, or receipt of chemotherapy for mCRPC. Patients/physicians planning treatment with chemotherapy during the 12 month period of the investigation are also ineligible.
* History of cognitive impairment or dysfunction, including a history of dementia, Alzheimer's disease, stroke with residual cognitive deficits, cognitive dysfunction related to alcohol or substance abuse, or cognitive dysfunction related to prior treatment for any cancer.
* Patients with a seizure history, history of recurrent falls, or known brain metastases are excluded from this clinical trial because of their poor prognosis and because of their heightened risk of seizure or progressive cognitive and/or neurologic dysfunction that would confound the evaluation.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III and IV heart failure), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations/substance abuse that would limit compliance with study requirements.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not eligible. Patients are not considered to have a "currently active" malignancy if they have completed all therapy and are now considered without evidence of disease for 1 year. Patients with cognitive dysfunction related to treatment of another malignancy, including a history of "chemo-brain", are ineligible.
* Patients taking psychotropic medications or illicit drugs that may alter cognition, concentration, or behavior. Appropriate treatment by a licensed provider with medications for depression or anxiety, including but not limited to SSRIs, SNRIs, and standard dose benzodiazepines at a stable dose, is permitted

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Cognitive function defined by overall Cogstate score and Cogstate module scores for each domain | Measured at baseline, 3 months, 6 months, and 12 months
  Raw scores on each module of the Cogstate test will be converted to standardized scores (z-scores and T-scores) according to age and/or education-adjusted published normative data per the Cogstate protocol. Linear regressions will be utilized to assess the mean differences between groups at each time point after the baseline while adjusting for baseline scores.

SECONDARY OUTCOMES:
Quality of life assessed using European Organization for Research and Treatment of Cancer quality of life questionnaire-C30 (EORTC QLQ C-30) | Measured at baseline, 3 months, 6 months, and 12 months
  The outcome measure for this questionnaire is the score as determined per standard scoring practices in the EORTC QLQ-C30 scoring manual. Mean scores from the EORTC QLQ-C30 survey instrument will be compared between groups at each time point, and changes in score will be assessed over time for each individual. Generalized linear regressions will be performed to estimate the differences between groups at each time point with adjustment for baseline and other covariates. GEE analysis will be used for the longitudinal data. Spearman p correlation coefficients between the standardized cognitive test scores and the mediators will be evaluated. Multivariable linear regressions for each time point will be performed to test the interactions between the group identity and each of the interested sociodemographic and clinical factors while adjusting for baseline and other covariates.
Fatigue assessed using Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT- Fatigue) | Measured at baseline, 3 months, 6 months, and 12 months
  The outcome measure for this questionnaire is the score as determined per standard scoring practices with the FACIT-Fatigue scoring manual. Mean scores from the FACIT-Fatigue survey instrument will be compared between groups at each time point, and changes in score will be assessed over time for each individual. Generalized linear regressions will be performed to estimate the differences between groups at each time point with adjustment for baseline and other covariates. GEE analysis will be used for the longitudinal data. Spearman p correlation coefficients between the standardized cognitive test scores and the mediators will be evaluated. Multivariable linear regressions for each time point will be performed to test the interactions between the group identity and each of the interested sociodemographic and clinical factors while adjusting for baseline and other covariates
Subjective measure of cognitive function by FACT-Cog | Measured at baseline, 3 months, 6 months, and 12 months
  The outcome measure for this questionnaire is the score as determined per standard scoring practices with the FACT-Cog scoring manual. Mean scores from the FACT-Cog survey instrument will be compared between groups at each time point, and changes in score will be assessed over time for each individual. Generalized linear regressions will be performed to estimate the differences between groups at each time point with adjustment for baseline and other covariates. GEE analysis will be used for the longitudinal data. Spearman p correlation coefficients between the standardized cognitive test scores and the mediators will be evaluated. Multivariable linear regressions for each time point will be performed to test the interactions between the group identity and each of the interested sociodemographic and clinical factors while adjusting for baseline and other covariates.
Depression by Patient Health Questionnaire (PHQ-9) | Measured at baseline, 3 months, 6 months, and 12 months
  The outcome measure for this questionnaire is the score as determined per standard scoring practices with the PH-Q 9 scoring manual. Mean scores from the PHQ-9 survey instrument will be compared between groups at each time point, and changes in score will be assessed over time for each individual. Generalized linear regressions will be performed to estimate the differences between groups at each time point with adjustment for baseline and other covariates. GEE analysis will be used for the longitudinal data. Spearman p correlation coefficients between the standardized cognitive test scores and the mediators will be evaluated. Multivariable linear regressions for each time point will be performed to test the interactions between the group identity and each of the interested sociodemographic and clinical factors while adjusting for baseline and other covariates.
Instrumental activities of daily living by Texas Functional Living Scale | Measured at baseline, 3 months, 6 months, and 12 months
  This measure will provide a score to represent patient's ability to complete daily tasks, and is a "direct assessment" based approach to measure instrumental activities of daily living.

OTHER OUTCOMES:
SNPs associated with cognitive function | SNP chip assessment using blood drawn at baseline or 3 month visit
  Multivariable linear regression will be utilized to compare the difference in primary outcomes between two allele groups at each time point for each SNP among patients in each treatment group. Baseline scores and other covariates will also be included in the model. Multivariable analyses using data from both treatment groups and control patients at each time point will be performed to identify SNPs whose associations with cognitive function are different between each treatment group and the control patients. The coefficient for the interaction between treatment group and allele group identity will be estimated and Wald-test p value will be provided. The p values will be ranked for the difference obtained from separate analysis for each SNP. A positive false discovery rate adjusted p values (q) will be calculated.
Imaging assessed by MRI | Baseline and 3 months
  MRI sequences will be compared by qualitative and quantitative analyses comparing MRI at baseline to MRI at 3 months for each patient. Changes will be compared qualitatively and quantitaively between treatment groups at baseline and 3 months also.

CONTACTS AND LOCATIONS:
Overall Officials: David VanderWeele, M.D., M.P.H., Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Tulane Cancer Center, New Orleans, Louisiana
  - University of Minnesota: Masonic Cancer Center, Minneapolis, Minnesota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided